CLINICAL TRIAL: NCT05895565
Title: A Phase 1b, Multicenter, Randomized, Double-blind, Placebo-controlled Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PMG1015 in Idiopathic Pulmonary Fibrosis (IPF) Subjects
Brief Title: A Multiple Ascending Doses (MAD) Study of PMG1015 in Idiopathic Pulmonary Fibrosis Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmongene Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMG1015_CHN_Ib
Record Dates: First submitted 2023-04-11; First posted 2023-06-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: IPF

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMG1015 (Experimental)
  Interventions: Drug: PMG1015
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: PMG1015 placebo

INTERVENTIONS:
Drug: PMG1015 — Including 3 dose levels: level 1, level 2 and level 3
  Arms: PMG1015
Drug: PMG1015 placebo — Including 2 dose levels corresponding to PMG1015 level 1 and level 2, with no placebo group set for PMG1015 level 3
  Arms: Placebo Comparator

SUMMARY:
This is a phase 1b randomized, double-blind, placebo-controlled, multiple ascending doses (MAD) study of PMG1015 in idiopathic pulmonary fibrosis (IPF) subjects. This study aims to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of PMG1015 after MAD.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of IPF as defined by current American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) Clinical Practice Guidelines for IPF (2022) (Pathological examination refers to transbronchial lung cryobiopsy or surgical/pleuroscopic lung biopsy);
2. Forced vital capacity percent predicted (FVCpp) ≥45% at screening;
3. Diffusing capacity of the lung for carbon monoxide (DLCO; corrected for haemoglobin) from 30% to 90% of the predicted, inclusive at screening;
4. Subjects not receiving any approved IPF treatment (pirfenidone or nintedanib) within 1 month before enrollment for any reasons

Key Exclusion Criteria:

1. Patients with instable condition of IPF as assessed by the investigator at screening, and those with acute exacerbation of IPF during screening or within 3 months prior to randomization;
2. Patients who are likely to be lung transplant recipients within 6 months or expected to survive less than 1 year as assessed by the investigator at screening;
3. Patients accompanying with an interstitial lung disease other than IPF;
4. Patients accompanying with other types of respiratory disorders, which may affect the study results as assessed by the investigator;
5. Patients who received vasodilator therapy for pulmonary arterial hypertension (e.g. Bosentan) within 1 month prior to screening;
6. Patients accompanying with other uncontrolled underlying diseases, for which the patient is not considered suitable for the study as assessed by the investigator;
7. Patients who had active tuberculosis within 12 months prior to screening, or clinical symptoms of bacterial, viral, fungal or microbial infections requiring intervention within 4 weeks prior to randomization;
8. Patients who have known allergic reaction to the investigational product or its active pharmaceutical ingredients (APIs), or history of allergic reaction to human, humanized, chimeric, or murine monoclonal antibodies or any substances contained in the excipients;
9. Pregnant or lactating women; female subjects who plan to become pregnant during the study, or patients who are not willing to take contraceptive measures as required by the protocol during the study;
10. Other conditions that preclude the patient from participating in the study as assessed by the investigator.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
The incidence of treatment-emergent adverse events (TEAEs) | Approximately 170 days.
  An Adverse Event (AE) is any event, side-effect or any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs are AEs that occur following the start of treatment.
The severity of treatment-emergent adverse events (TEAEs) | Approximately 170 days.
  Severity of TEAEs (Grade 1 to 5) will be assessed based on NCI-CTCAE V5.0.
The incidence of serious adverse events (SAEs) | Approximately 170 days.
  A serious adverse event (SAE) is defined as an AE occurring during any study phase and at any dose of medicinal product that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, or results in congenital anomaly/birth defect.
The severity of serious adverse events (SAEs) | Approximately 170 days.
  A serious adverse event (SAE) is defined as an AE occurring during any study phase and at any dose of medicinal product that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, or results in congenital anomaly/birth defect.
Assessment of pulmonary function test results-forced vital capacity (FVC) | Approximately 170 days.
  Pulmonary function test is a test to explore the functional status of human respiratory system with the knowledge of exercise respiratory physiology and modern examination technology. Forced vital capacity (FVC) (mL) will be measured at Visits 1, 8, 14 and 16, to assess the changes in FVC from baseline to post-dose.
Assessment of pulmonary function test results-forced vital capacity percent predicted (FVCpp) | Approximately 170 days.
  Pulmonary function test is a test to explore the functional status of human respiratory system with the knowledge of exercise respiratory physiology and modern examination technology. Forced vital capacity percent predicted (FVCpp) (%) will be measured at Visits 1, 8, 14 and 16, to assess the changes in FVCpp from baseline to post-dose.
Assessment of pulmonary function test results-forced expiratory volume in 1 second (FEV1) | Approximately 170 days.
  Pulmonary function test is a test to explore the functional status of human respiratory system with the knowledge of exercise respiratory physiology and modern examination technology. Forced expiratory volume in 1 second (FEV1) (L) will be measured at Visits 1, 8, 14 and 16, to assess the changes in FEV1 from baseline to post-dose.
Assessment of pulmonary function test results-diffusing capacity of the lungs for carbon monoxide (DLCO) | Approximately 170 days.
  Pulmonary function test is a test to explore the functional status of human respiratory system with the knowledge of exercise respiratory physiology and modern examination technology. Diffusing capacity of the lungs for carbon monoxide (DLCO) (mL/min/mmHg) will be measured at Visits 1, 8, 14 and 16, to assess the changes in DLCO from baseline to post-dose.
Assessment of pulmonary function test results-diffusing capacity of the lungs for carbon monoxide percent predicted (DLCOpp) | Approximately 170 days.
  Pulmonary function test is a test to explore the functional status of human respiratory system with the knowledge of exercise respiratory physiology and modern examination technology. Diffusing capacity of the lungs for carbon monoxide percent predicted (DLCOpp) (DLCO%) will be measured at Visits 1, 8, 14 and 16, to assess the changes in DLCOpp from baseline to post-dose.

SECONDARY OUTCOMES:
Evaluate the area under the serum drug concentration-time curve from time zero to the last quantifiable time point (AUC0-t) of PMG1015. | Approximately 170 days.
  AUC is a pharmacokinetic parameter that represents the concentration of a drug in the blood at a certain time.
Evaluate the area under the serum drug concentration-time curve from time zero to infinity (AUC0-∞) of PMG1015. | Approximately 170 days.
  AUC is a pharmacokinetic parameter that represents the concentration of a drug in the blood at a certain time.
Evaluate the area under the concentration-time curve from time zero to the end of a dosing interval (AUC0-tau) of PMG1015. | Approximately 170 days.
  AUC is a pharmacokinetic parameter that represents the concentration of a drug in the blood at a certain time.
Evaluate the maximum concentration (Cmax) of PMG1015. | Approximately 170 days.
  Cmax refers to the highest concentration of a drug in the blood after administration, which is related to the dose, route of administration, dosing frequency, and time to reach the peak concentration.
Evaluate the time to reach the maximum concentration (Tmax) of PMG1015. | Approximately 170 days.
  Tmax refers to the time when a drug reaches its maximum concentration and exhibits its maximum effect in the body.
Evaluate the half-life (t1/2) of PMG1015. | Approximately 170 days.
  t1/2 refers to the time required for the drug concentration in the blood to decrease by half.
Evaluate the clearance rate (CL) of PMG1015. | Approximately 170 days.
  CL is the volume of blood that is completely cleared of a drug per unit time by the excretory organs, and its unit is usually mL·(min·kg)-1 or L·(h·kg)-1.
Evaluate the distribution volume (Vz) of PMG1015. | Approximately 170 days.
  Vz is a pharmacokinetic parameter that reflects the extent of drug distribution in various tissues in the body.
Evaluate the elimination rate constant (λz) of PMG1015. | Approximately 170 days.
  λz is referred to as the elimination rate constant, which is defined as the ratio of the amount of compound eliminated per unit time to the total amount, with its unit being the reciprocal of time.
Correlation between the dose and exposure. | Approximately 170 days.
  Dose refers to the quantity of drug administered at one time to achieve the desired therapeutic effect, and it can vary depending on the patient's needs and medical condition.
Incidence of PMG1015-induced and PMG1015-boosted ADAs. | Approximately 170 days.
  Immunogenicity assessment is mainly based on anti-drug antibodies (ADAs), including the incidence of PMG1015-induced and PMG1015-boosted ADAs.

CONTACTS AND LOCATIONS:
Overall Officials: Wang, Principal Investigator — China-Japan Friendship Hospital; Dai, Principal Investigator — China-Japan Friendship Hospital
Locations (7):
- China (7):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Tongji Hospital Tongji Medical College of HUST, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No